CLINICAL TRIAL: NCT01219920
Title: Phase III Trial of Infusional Fluorouracil, Leucovorin, Oxaliplatin and Irinotecan (FOLFOXIRI) Compared With Infusional Fluorouracil, Leucovorin and Irinotecan (FOLFIRI) as First-line Treatment for Metastatic Colorectal Cancer
Brief Title: FOLFOXIRI Compared With FOLFIRI for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASL601LIOM03; 2007-002886-11 (EudraCT Number)
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; Phase III; FOLFOXIRI; FOLFIRI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — IFL protocol; Irinotecan; Fluorouracil; FOLFOXIRI protocol; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFIRI (Active Comparator): Irinotecan 180 mg/sqm on day 1 Leucovorin 100 mg/sqm on day 1 and day 2 5-fluorouracil 400 mg/sqm bolus followed by 5-fluorouracil 600 mg/sqm 22-hour continuous infusion on day 1 and day 2 Repeated every 2 weeks
  Interventions: Drug: FOLFIRI
- FOLFOXIRI (Experimental): Irinotecan 165 mg/sqm on day 1 Oxaliplatin 85 mg/sqm on day 1 Leucovorin 200 mg/sqm on day 1 5-fluorouracil 3200 mg/sqm 48-hour continuous infusion starting on day 1 Repeated every 2 weeks
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFIRI — Irinotecan 180 mg/sqm on day 1 Leucovorin 100 mg/sqm on day 1 and day 2 5-fluorouracil 400 mg/sqm bolus followed by 5-fluorouracil 600 mg/sqm 22-hour continuous infusion on day 1 and day 2 Repeated every 2 weeks
  Other Names: Campto; l-lederfolin; 5-FU
  Arms: FOLFIRI
Drug: FOLFOXIRI — Irinotecan 165 mg/sqm on day 1 Oxaliplatin 85 mg/sqm on day 1 Leucovorin 200 mg/sqm on day 1 5-fluorouracil 3200 mg/sqm 48-hour continuous infusion starting on day 1 Repeated every 2 weeks
  Other Names: Campto; Eloxatin; l-leucovorin; 5FU
  Arms: FOLFOXIRI

SUMMARY:
The purpose of the study is to evaluate if the exposure to all the three active cytotoxic agents (FOLFOXIRI regimen) is superior in terms of response rate to conventional chemotherapy with the FOLFIRI regimen as first-line treatment of metastatic colorectal cancer patients.

DETAILED DESCRIPTION:
Survival of patients with metastatic colorectal cancer is correlated with the proportion of patients who receive all the three active drugs in the course of the disease, but not with the proportion of patients who receive any second-line therapy. In a sequential strategy, not all patients who progress after first-line chemotherapy are able to receive second-line treatment. Moreover, there is a correlation between the response rate to chemotherapy and the postchemotherapy radical resection rate of metastases.

Therefore, a way to improve the outcome of metastatic colorectal cancer patients could be to administer a first-line regimen containing the three active agents.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of the colon or rectum
* unresectable metastatic disease
* age 18 to 75 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or lower if age 70 years or younger or ECOG performance status of 0 if age 71 to 75 years measurable disease according to WHOcriteria
* leukocyte count of at least 3,500/mm3, neutrophils count of at least 1,500/mm3, platelet count of at least 100,000/mm3
* serum creatinine of 1.3 mg/dL or less
* serum bilirubin less than 1.5 mg/dL and AST, ALT, and alkaline phosphatase 2.5 x normal values or less (</= 5 if liver metastases)
* previous fluoropyrimidine-based adjuvant chemotherapy was allowed if ended more than 6 months before random assignment

Exclusion Criteria:

* previous palliative chemotherapy for metastatic disease
* previous chemotherapy including irinotecan or oxaliplatin
* symptomatic cardiac disease, myocardial infarction in the last 24 months or uncontrolled arrhythmia
* active infections
* inflammatory bowel disease
* total colectomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2001-11; Primary Completion 2005-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) | Responses are evaluated every 8 weeks according to WHO criteria and reviewed by an independent panel at the end of treatment (6 months)
  Responses are evaluated every 8 weeks according to WHO criteria. The determination of responses and progression was initially based on investigator-reported measurements; computed tomography scans of all responding patients and of patients with stable disease were subsequently subjected to external review by an independent panel.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Progressions are evaluated every 8 weeks according to WHO criteria and reviewed by an independent panel at the end of follow up (36 months)
  PFS is defined as the length of time from random assignment to disease progression or to death resulting from any cause, whichever occurred first, or to last contact.
Overall survival (OS) | For survival analysis participants are followed until death
  OS is defined as the length of time from random assignment to death or to last contact.
Postchemotherapy radical (R0) surgical resection rate of metastases | Postchemotherapy radical (R0) surgical resection rate of metastases were evaluated every 8 weeks during treatment and during follow up (36 months)
  Percentage of patients who undergo radical (R0) resection of metastases after achieving objective response to chemotherapy.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Number of Participants with Adverse Events as a Measure of Safety and Tolerability were evaluated every 2 weeks during treatment and every 8 weeks during follow up (36 months)
  During the full lenght of first-line treatment, number of enrolled patients reporting adverse events is recorded. Adverse events are evaluated according to National Cancer Institute Common Toxicity Criteria version 2.0.
Quality of life (QoL) | Quality of life was evaluated every 2 weeks during treatment and every 8 weeks during follow up (36 months)
  Quality of life is assessed at the beginning of each treatment cycle using the Quality of Life Questionnaire of the European Organisation for Research and Treatment of Cancer (version 2.0).
  The QLQ-C30 questionnaire was analyzed with the global health status/quality-of-life scale as the primary end point and the other 10 scales as secondary end points.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Falcone, MD, Principal Investigator — University of Pisa
Locations (48):
- Italy (48):
  - Ospedale Civile Ss. Antonio E Biagio Di Alessandria - Alessandria (Al) Oncologia Medica, Alessandria
  - A.O. Universitaria Ospedali Riuniti - Ospedale Umberto I Di Ancona - Ancona (An) Oncologia Medica, Ancona
  - Ausl Della Valle D' Aosta (Ao) - Aosta (Ao) Oncologia Medica, Aosta
  - P.O. Zona Aretina - Ospedale S. Donato Di Arezzo - Arezzo (Ar) Oncologia Medica, Arezzo
  - Azienda Ospedale 'G.Rummo' - Benevento (Bn) Oncologia Medica, Benevento
  - Ospedale Degli Infermi Di Biella - Biella (Bi) Oncologia Medica, Biella
  - Ospedale S. Orsola F.B.F. - Brescia - Brescia (Bs) Oncologia Medica, Brescia
  - Stabilimento "Perrino" - Brindisi - Brindisi (Br) Oncologia Medica, Brindisi
  - Azienda Ospedaliera S. Elia - Caltanissetta (Cl) Oncologia Medica, Caltanissetta
  - Ospedale Versilia - Camaiore (Lu) Oncologia Medica, Camaiore
  - Ospedale Cecina - Cecina (Li) Oncologia Medica, Cecina
  - Istituti Ospitalieri - Cremona - Cremona (Cr) Oncologia Medica, Cremona
  - Azienda Ospedaliera S. Croce E Carle Di Cuneo - Cuneo (Cn) Oncologia Medica, Cuneo
  - Ausl 11 Di Empoli (Fi) - Empoli (Fi) Oncologia Medica, Empoli
  - Asur - Zona Territoriale 6 Di Fabriano (An) - Fabriano (An) Oncologia Medica, Fabriano
  - Ospedale Santa Croce Fano - Fano (Pu) Oncologia Medica, Fano
  - Ausl 10 Di Firenze - Firenze (Fi) Oncologia Medica, Florence
  - A.O. Universitaria Careggi Di Firenze Oncologia Medica, Florence
  - E.O. Ospedali Galliera - Genova (Ge) Oncologia Medica, Genova
  - Irccs Istituto Nazionale Per La Ricerca Sul Cancro (Ist) - Genova (Ge) Oncologia Medica, Genova
  - Ospedale Sant'Andrea La Spezia - La Spezia (Sp) Oncologia Medica, La Spezia
  - Ausl Le Di Lecce - Lecce (Le) Oncologia Chirurgica, Lecce
  - Ospedale Per Acuti "Mater Salutis" Legn. - Legnago (Vr) Oncologia Medica, Legnano
  - U.O. Oncologia Medica, Ospedale Civile, Livorno
  - Presidio Ospedaliero Piana Di Lucca - Lucca (Lu) Oncologia Medica, Lucca
  - Irccs Fondazione Centro S. Raffaele Del Monte Tabor - Milano (Mi) Oncologia Medica, Milan
  - Ospedale Ca' Granda-Niguarda - Milano - Milano (Mi) Oncologia Medica, Milan
  - Ospedale Civile Di Mirano - Mirano (Ve) Oncologia Medica, Mirano
  - A.O. Universitaria Federico Ii Di Napoli Oncologia Medica, Napoli
  - A.O. Universitaria Maggiore Della Carita' Di Novara Oncologia Medica, Novara
  - A.O. Universitaria Di Parma Oncologia Medica, Parma
  - Asl 1 Di Citta' Di Castello (Pg) - Citta' Di Castello (Pg) Oncologia Medica, Perugia
  - A.O. Di Perugia - Ospedale S. Maria Della Misericordia (Ex Silvestrini) - Perugia (Pg) Oncologia Medica, Perugia
  - Azienda Ospedaliera San Salvatore - Pesaro (Pu) Oncologia Medica, Pesaro
  - Ospedale Piombino - Piombino (Li) Oncologia Medica, Piombino
  - Ausl 5 Di Pisa - Pisa (Pi) Oncologia Medica, Pisa
  - A.O. Universitaria Pisana - Pisa (Pi) Oncologia Medica, Pisa
  - A.O. Universitaria Pisana Oncologia Medica, Pisa
  - Ausl 3 Di Pistoia - Pistoia (Pt) Oncologia Medica, Pistoia
  - Ospedali Riuniti Di Pistoia - Pistoia (Pt) Oncologia Medica, Pistoia
  - Ospedale Di S. Maria Nuova - Reggio Nell'Emilia, Reggio Emilia
  - Policlinico Universitario Campus Bio-Medico Di Roma Oncologia Medica, Roma
  - Policlinico Umberto I Di Roma Oncologia Medica, Roma
  - Policlinico Universitario Gemelli Di Roma Oncologia Medica, Roma
  - A.O. Universitaria Senese Oncologia Medica, Siena
  - Ausl 7 Di Siena - Siena (Si) Oncologia Medica, Siena
  - Ospedale Civile - Sondrio - Sondrio (So) Oncologia Medica, Sondrio
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino Oncologia Medica, Torino

REFERENCES:
- [Background] Falcone A, Ricci S, Brunetti I, Pfanner E, Allegrini G, Barbara C, Crino L, Benedetti G, Evangelista W, Fanchini L, Cortesi E, Picone V, Vitello S, Chiara S, Granetto C, Porcile G, Fioretto L, Orlandini C, Andreuccetti M, Masi G; Gruppo Oncologico Nord Ovest. Phase III trial of infusional fluorouracil, leucovorin, oxaliplatin, and irinotecan (FOLFOXIRI) compared with infusional fluorouracil, leucovorin, and irinotecan (FOLFIRI) as first-line treatment for metastatic colorectal cancer: the Gruppo Oncologico Nord Ovest. J Clin Oncol. 2007 May 1;25(13):1670-6. doi: 10.1200/JCO.2006.09.0928. PMID 17470860
- [Background] Masi G, Vasile E, Loupakis F, Bursi S, Ricci S, Petrini I, Fontana A, Allegrini G, Falcone A. Triplet combination of fluoropyrimidines, oxaliplatin, and irinotecan in the first-line treatment of metastatic colorectal cancer. Clin Colorectal Cancer. 2008 Jan;7(1):7-14. doi: 10.3816/CCC.2008.n.002. PMID 18279572
- [Background] Masi G, Loupakis F, Pollina L, Vasile E, Cupini S, Ricci S, Brunetti IM, Ferraldeschi R, Naso G, Filipponi F, Pietrabissa A, Goletti O, Baldi G, Fornaro L, Andreuccetti M, Falcone A. Long-term outcome of initially unresectable metastatic colorectal cancer patients treated with 5-fluorouracil/leucovorin, oxaliplatin, and irinotecan (FOLFOXIRI) followed by radical surgery of metastases. Ann Surg. 2009 Mar;249(3):420-5. doi: 10.1097/SLA.0b013e31819a0486. PMID 19247029
- [Derived] Cremolini C, Loupakis F, Masi G, Lonardi S, Granetto C, Mancini ML, Chiara S, Moretto R, Rossini D, Vitello S, Allegrini G, Tonini G, Bergamo F, Tomasello G, Ronzoni M, Buonadonna A, Bustreo S, Barbara C, Boni L, Falcone A. FOLFOXIRI or FOLFOXIRI plus bevacizumab as first-line treatment of metastatic colorectal cancer: a propensity score-adjusted analysis from two randomized clinical trials. Ann Oncol. 2016 May;27(5):843-9. doi: 10.1093/annonc/mdw052. Epub 2016 Feb 9. PMID 26861604